CLINICAL TRIAL: NCT05039385
Title: Impact of a Supervised Physical Exercise Program (ESATRAL) in Patients With Anorexia Nervosa After Hospital Discharge
Brief Title: Exercise Program in Patients With Anorexia Nervosa (ESATRAL)
Acronym: ESATRAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough sample was obtained
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Collaborators: PERFORMA Salud S.L. (Unknown); ITA PREVI Valencia (Unknown)
Responsible Party: Principal Investigator, Ana Pablos Monzó, Principal investigator, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2019-2020/143
Record Dates: First submitted 2021-07-22; First posted 2021-09-09 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Anorexia
Keywords: Exercise; Resistance training; Anorexia; Physical activity; Anorexia nervosa; Eating disorders; Exercise treatment
MeSH Terms: conditions — Anorexia; Motor Activity; Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This project is based on an, longitudinal, prospective, controlled, randomized, intervention study and blind for the researchers responsible for the study. Thus, the subjects participating in the study will be divided into 2 groups, one of which will perform the exercise program (intervention group, IG), and another that will follow their daily routine treatment without added exercise (control group, CG).
  Each group will have 4 measurements in which the corresponding variables will be evaluated: A) before the start of the intervention, B) at 3 months (12 weeks), C) at 6 months (at the end of the intervention, 24 weeks), D) at 9 months (3 months post-intervention, 36 weeks).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator: The persons who make the data analysis and decide whether a patient has experienced an outcome of interest will be masked.
  Outcome assessors: The persons who assess patients and provide outcome data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESATRAL Group (Experimental): They will perform the supervised physical exercise program. The supervised exercise program (ESATRAL) will last 24 weeks with 2-3 non-consecutive weekly sessions. The duration of each session will be 30 minutes and will progressively increase depending on the phase in which we are until reaching 60 minutes.
  Interventions: Other: Exercise Program focused on resistance training
- Control Group (No Intervention): They will follow their daily treatment without added exercise

INTERVENTIONS:
Other: Exercise Program focused on resistance training — The program will be carried out by a personal trainer. To ensure correct execution, given that the groups will be of a maximum of 5 people. Each session will include:
  A) Warm up: movility exercises and coordination games B) Main part: 3 exercises will be included to strengthen different muscle groups (pull , bench press and back squat). Velocity based training (VBT) will be used to control load. 3 sets of 16-30 repetitions mantaining the speed between Light (estimated loss of speed of the series 5-10%).
  C) Cool down: feedback with patients based on the work of Stiles-Shields (2015).
  Specific training content will focus on safety, while re-educating patients on proper exercise methods, motivation-related attitudes, and transparency on health benefits and potential harms as a result of increased exercise.
  Arms: ESATRAL Group

SUMMARY:
Excessive physical exercise is one of the main symptoms of anorexia and a common restrictive behavior used by patients, which is associated with less short- and long-term treatment success. Supervised exercise has shown these benefits in patients with anorexia: opportunity to learn and acquire knowledge and information on how to perform physical activity in a healthy, safe and moderate way, less feelings of incapacity; lower risk of relapse; prohibiting exercise during treatment can increase the likelihood that patients will revert to old patterns once therapy is completed. Exercise can be as effective as antidepressants and psychological therapies to treat some cases of depression present in anorexia.

The objective of the ESATRAL program is to analyze the physiological, psychological, body composition, physical condition and functionality effects of a supervised strength-focused training program in patients with anorexia nervosa after hospital discharge. All participants are assessed at baseline, after 12 weeks, post-treatment (24 weeks), and at 9 months' post follow-up (36 weeks).

DETAILED DESCRIPTION:
Experts in eating disorders recommend restricting exercise until the person is medically stable, of sufficient weight and able to compensate exercise with sufficient energy intake. In this sense, a reintroduction and promotion of healthy exercise should be done in a graded and supervised manner, where exercise would provide great benefits, such as improving social confidence and providing a tool for healthy living. That is the goal of the ESATRAL (EXCERCISE AND HEALTH IN EATING DISSORDERS) program. The relationship between eating disorders (ED) and exercise has been controversial, but different studies have already shown that the therapeutic use of exercise in the treatment could be positive if used as a tool for healthy living. Historically in the literature, exercise in anorexia has been mainly considered as a problematic activity that should be limited or even completely forbidden, especially during the acute phase of the disorder, but different researchers have already questioned the restriction-based approach to exercise and investigated its potentially healthy role in recovery. It should also be noted that restricting physical activity can have detrimental musculoskeletal and cardiometabolic consequences for patients with anorexia. In addition to experiencing significant strength losses and atrophy of type II muscle fibers, the loss of lean tissue affects organ mass and function in these patients. Lean body mass-comprised of visceral organs such as the liver and heart, as well as bone and skeletal muscle-plays an important role in setting the demand for energy metabolism. Patients with anorexia present with a number of characteristic metabolic and endocrine disorders as a result of chronic malnutrition that affect lean tissue. ESATRAL is a supervised physical exercise program that is implemented in patients with anorexia nervosa after hospital discharge. ESATRAL consists of three days of weekly strength training that will be measured following the strength-velocity methodology. The objective of the ESATRAL program is to analyze the physiological, psychological, body composition, physical condition and functionality effects of a supervised strength-focused training program (6 month duration) in patients with anorexia nervosa after hospital discharge. The risk of relapse is an obstacle that can be minimized if supervised exercise were included in the treatment of anorexia as is done in ESATRAL. Many patients engage in excessive and unsupervised exercise, and returning to this level of physical activity after treatment has been associated with an increased risk of relapse. Therefore, prohibiting exercise during treatment may increase the likelihood that patients will fall back into old patterns after treatment ends, hence the importance of ESATRAL.

The ESATRAL project will compare the effects of supervised strength training as a part of the treatment vs. treatment without supervised strength training, in patients with Anorexia nervosa after hospital discharge. All participants will be assessed at baseline, after 12 weeks, post-treatment (24 weeks), and at 9 months' post follow-up (36 weeks). .

The study will be conducted with ITA- PREVI patients at the PERFORMA personal training health center in Valencia.

ELIGIBILITY:
Inclusion Criteria:

* Women with a BMI higher than 15 Kg / m2,
* aged between 16 to 45 years old,
* diagnosed with restrictive (DSM-V F50.01) or purgative (F50.02 (DSM-V) anorexia.
* Patients from the 24 h or Day Hospital and ambulatory.
* who has agreed to participate in the study and signed the informed consent or in case of being minors, their father / mother / legal guardian signs the participation consent.

Exclusion Criteria:

* Patients with contraindication in the performance of physical exercise (cardiovascular risk factors),
* patients with severe mental disorder (major depressive episode, bipolar disorder, severe personality disorders, schizophrenia)
* Patients who refuse to sign the informed consent.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Risk of eating disorders | Base line, week 12, week 24, week 36
  The Eating Disorder Inventory-3 will be used. It made up of 91 items organized into 12 subscales (3 specific to eating disorders and 9 general psychological scales). It uses a 0-4 point scoring system. Higher scores indicating greater risk of an eating disorder.
Changes in Maximal strength horizontal pull based on the execution velocity. | Base line, week 12, week 24, week 36
  Difference in muscle strength measured with horizontal pull strength tests in patients treated with standard treatment compared to patients treated with ESATRAL. To measure muscle strength we will use a linear encoder (T-FORCE dynamic measurement system) to achieve the movement speed. The exercise will be done in a Smith Machine.
Changes in Maximal strength bench press based on the execution velocity. | Base line, week 12, week 24, week 36
  Difference in muscle strength measured with horizontal bench press tests in patients treated with standard treatment compared to patients treated with ESATRAL. To measure muscle strength we will use a linear encoder (T-FORCE dynamic measurement system) to achieve the movement speed. The exercise will be done in a Smith Machine.
Changes in Maximal strength squat based on the execution velocity. | Base line, week 12, week 24, week 36
  Difference in muscle strength measured with squat tests in patients treated with standard treatment compared to patients treated with ESATRAL. To measure muscle strength we will use a linear encoder (T-FORCE dynamic measurement system) to achieve the movement speed. The exercise will be done in a Smith Machine.

SECONDARY OUTCOMES:
Changes in Blood pressure | Base line, week 12, week 24, week 36
  Changes related to blood pressure (systolic and diastolic pressure) will be measured in patients treated with standard treatment compared to patients treated with ESATRAL with an Omron Digital Automatic Blood Pressure Monitor Hem Arm 7114 with pediatric cuff (mmHg).
Changes in Bone Mineral Density | Base line, week 24, week 36
  Difference in bone mineral density (BMD) measured by Dual-energy X-ray Absorptiometry (DXA) (total bone mineral content, BMD lumbar spine and femur neck) in patients treated with standard treatment compared to patients treated with ESATRAL. It will be measured in g/m2].
Changes in Heart Rate | Base line, week 12, week 24, week 36
  Difference in heart rate measured with Polar RS800CX heart rate monitor in patients treated with standard treatment compared to patients treated with ESATRAL (beats per minute).
Restoration of ovarian function | Base line, week 12, week 24, week 36
  Changes in ovarian function from interviews conducted by the endocrine physician in patients treated with standard treatment compared to patients treated with ESATRAL (answer: yes, no).
Changes in Height | Base line, week 12, week 24, week 36
  It will be measured by attaching a Seca scale to the Seca 714 scale (Seca Vogel & Halke GmbH & Co. KG, Hamburg, Germany), with an accuracy of 0.1 cm.
Changes in bodyweight | Base line, week 12, week 24, week 36
  Difference in bodyweight (kg) with Tanita MC-780MA in patients treated with standard treatment compared to patients treated with ESATRAL.
Changes in corporal composition | Base line, week 12, week 24, week 36
  Difference in fat mass (kg), and fat free mass (kg) measured with DXA and Tanita MC-780MA in patients treated with standard treatment compared to patients treated with ESATRAL.
Demographic variables | Base line, week 12, week 24, week 36
  The following demographic variables will be taken to characterize the sample:
  Age, type of anorexia (diagnosed in the Hospital), time of evolution of the disease and BMI (BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared).
Changes in perceived quality of life | Base line, week 12, week 24, week 36
  Difference in quality of life measured with SF-12v2 (Ware et al., 2009) in patients treated with standard treatment compared to patients treated with ESATRAL. Scoring is on a scale from 0 to 100 where higher score means a better perceived state of health.
Changes in eating attitudes | Base line, week 12, week 24, week 36
  Difference in attitudes towards food measured with EAT-26 (Garner et al., 1982) in patients treated with standard treatment compared to patients treated with ESATRAL.
  Scoring is on a scale from 0 to 78. Higher scores indicate greater risk of an eating disorder and total scores 20 or above are considered to be in the clinical range.
Changes in compulsive exercise | Base line, week 12, week 24, week 36
  Difference in compulsive exercise measured with Compulsive Exercise test (CET) in patients treated with standard treatment compared to patients treated with ESATRAL. Scoring is measured on a scale from 0 to 5 where higher score means a worse outcome except for two questions where higher score means better outcome.
Changes in body image | Base line, week 12, week 24, week 36
  Difference in body image measured through the Multidimensional Body Self Relations Questionnaire (MBSRQ) (Cash, 2000) in patients treated with standard treatment compared to patients treated with ESATRAL. Scoring is measured on a scale from 0 to 5 where the higher the score, the greater the satisfaction with one's own body image.
Changes in agility | Base line, week 12, week 24, week 36
  Difference in agility measured with the 3 and 10 m Time Up and Go (TUG) test (San Juan et al. 2008) and the Timed Up and Down Stairs (TUDS) test (Gocha et al. 2001) in patients treated with standard treatment compared to patients treated with ESATRAL. In both tests the time necessary to perform the test is taken and the longer the time the worse the agility.
Structured physical activity | Base line, week 12, week 24, week 36
  Daily time spent in structured ligth, moderate or vigorous intensity (percentage) physical activity will be measured using the ActiGraph GT9X Link to compare patients treated with standard treatment with patients treated with ESATRAL.
Changes in physical performance of the lower extremities | Base line, week 12, week 24, week 36
  Difference in the physical performance of the lower extremities measured with the Short Physical Performance Battery in patients treated with standard treatment compared to patients treated with ESATRAL.
Changes in functionality | Base line, week 12, week 24, week 36
  Difference in the function of the participants with respect to day-to-day activities measured with the Barthel Index (Mahoney and Barthel, 1965) in patients treated with standard treatment compared to patients treated with ESATRAL. The range of scores obtained goes from 0 to100 points. A total score of 100 indicates complete self-sufficiency in performance, while a score of zero would indicate absolute dependence. A score obtained between 21 and 60 is indicative of a severe dependency, while scores higher than this limit of 60 points would describe almost all the people who are independent for the execution of these activities.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Pablos Monzo, PhD, Principal Investigator — Catholic University of Valencia
Locations (1):
- Ita Previ Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers